CLINICAL TRIAL: NCT02886663
Title: Visual Field Restoration in Patients With Post-stroke Homonymous Hemianopsia
Acronym: REVOIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major inclusion difficulties
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OGT_2015_16
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hemianopsia
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate rehabilitation (Experimental)
  Interventions: Other: stimulation of the blind visual field
- delayed rehabilitation (Other)
  Interventions: Other: stimulation of the blind visual field

INTERVENTIONS:
Other: stimulation of the blind visual field

SUMMARY:
This study will assess the effectiveness of a stimulus, in the blind field of hemianopsic patients, to restore the vision of patients with homonymous hemianopsia consecutive to stroke (unilateral occipital lesion). Hemianopsia occurs in 30% of strokes regardless of the cerebral localization and in 60% of stroke interesting the territory of the posterior cerebral artery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an homonymous visual field amputation after vascular retrochiasmatic lesion of the occipital region (visual cortex alone or with optical radiations or with other associated occipital areas)
* inclusion 3 months to 36 months after stroke
* Patients aged 18 years and older

Exclusion criteria:

* Brain injury history
* Severe neuropsychological, psychiatric or behavioral disorder
* Severe eye disorder or visual impairment (visual acuity less than 3/10)
* Progressive eye disorder (cataracts or glaucoma)
* insufficient French language proficiency to understand the questionnaires and rehabilitation tasks
* patient under legal protection
* patient's opposition to participate in the study
* no medical insurance coverage
* pregnant pr breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
change in the sensitivity of detection of a visual stimulus after rehabilitation | change from baseline sensitivity at week 22
  change in the mean number of points where the sensitivity is lower than 15db in each contralesional hemifield, before and after rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie CHOKRON, Study Director — Fondation OPH A de Rothschild; Olivier GOUT, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France